CLINICAL TRIAL: NCT05745415
Title: Cancer Stem Cell Specific Aptamer's Ability to Detect Blood Circulating Cancer Stem Cells and Its Role as a Predictor of Prognosis in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-1161
Record Dates: First submitted 2023-01-29; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An aptamer is a single-stranded nucleic acid (DNA, RNA) that has a stable tertiary structure and binds to a target molecule with high binding force and specificity. To determine the prognosis of pancreatic cancer through cancer stem cell-specific aptamer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreatic cancer patients

SUMMARY:
The treatment performance of pancreatic cancer has not changed significantly over the past 20 years and is still less than 10%. In addition, 80-90% of pancreatic cancer patients are found to be already advanced at the time of diagnosis, and it is the best malignant tumor in the human body with a 5-year survival rate of less than 10% and a median survival period of less than 1 year. However, early diagnosis of pancreatic cancer is still difficult, and there is no effective treatment other than surgery, so the increase in long-term survival rate over the past 20 years has been insignificant or stagnant. The response rate to anticancer drug treatment after surgery or anticancer drug when surgery is not possible is only around 20%, so it is very urgent to discover new biomarkers in predicting drug resistance and recurrence after surgery and predicting prognosis in advance. Minimally non-invasive diagnostic techniques are very important to detect and track cancer progression in the clinic. In particular, histological diagnosis and analysis have limitations in carcinomas, such as pancreatic cancer, which are small and distant, making it difficult to obtain tissue samples. CA 19-9, a prognostic marker for existing pancreatic cancer, 1) has low specificity for early diagnosis of pancreas, 2) is not detected in lewis A, B antibody-negative patients, and 3) shows false positive in cases with cholangitis at the same time. Because it has many disadvantages, the development of prognostic biomarkers in blood is urgently needed.

Recently, a study has been reported that the presence or absence of detection of circulating tumor cells is directly related to the prognosis of pancreatic cancer patients, and can be used for monitoring the patient's treatment response and for recurrence after surgery. In particular, the process of cancer metastasis consists of epithelial-to-mesenchymal transition and migration of cancer cells into the blood, and the existence of cancer stem cells is very important for metastasis and drug treatment resistance. Eventually, it is known to cause pancreatic cancer metastasis and recurrence.

Cancer stem cells have the ability to self-renew, the capability of developing, multiple cell lineages, and the potential of extensive proliferation, and the ability to detect cancer stem cells in the blood is important in pancreatic cancer patients who are at high risk of metastasis and recurrence. It is a non-invasive screening tool. Comparatively evaluate the treatment response and prognosis of pancreatic cancer patients according to the characteristics and subtypes of circulating cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 20 years of age
* Patients diagnosed with pancreatic cancer histologically or radiologically

Exclusion Criteria:

* non-pancreatic cancer
* Patients who failed to obtain informed consent from the patient

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 20 who have been diagnosed with pancreatic cancer histologically or radiologically.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Progression free survival | the duration from treatment initiation to disease progression (Up to 100 weeks)
  Progression free survival : The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Overall survival | he duration from diagnosis of pancreatic cancer to death or last follow-up (up to 100 weeks)
  Overall survival : The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Si Young Song, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea